CLINICAL TRIAL: NCT00354471
Title: Short and Long Term Outcomes of Uterine Artery Embolization.
Brief Title: Uterine Artery Embolization for Symptomatic Fibroids
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Other Study IDs: B2000 115
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2006-07

CONDITIONS: Uterine Fibroids; Menorrhagia; Adenomyosis
MeSH Terms: conditions — Leiomyoma; Menorrhagia; Adenomyosis | interventions — Uterine Artery Embolization

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Uterine Artery Embolization

SUMMARY:
This study will evaluate the safety, efficacy , quality of life and patient satisfaction of uterine artery embolization for the treatment of symptomatic uterine fibroids. It will provide useful information in the development od guidelines in patient selection, procedural management and subsequent follow up.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms related to the pressence of uterine fibroids serious enough to consider surgical options
* Confirmation of fibroids by endovaginal and transabdominal ultrasound

Exclusion Criteria:

* Pedunculated fibroids
* Desire for fertility
* Carcinoma of pelvic organs
* Previous pelvic irradiation
* Bleeding diathesis and vasculitis
* History of allergiy to contrst medium

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Boroditsky, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada